CLINICAL TRIAL: NCT04391400
Title: The Use of Peripheral Blood Specimens From Patients Suspected of Having SARS-CoV-2 Infections in Research Studies Intended to Support the Development of COVID-19 Detection Methods, Treatments, and/or Vaccines
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Invivoscribe, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IVS-000-002
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The donated specimens will be:
  * From patients suspected of SARS-CoV-2 viral infections.
  * At least 2mL to 5mL of peripheral blood.
  * Collected in EDTA tubes.
  * Shipped to ambient LabPMM, LLC within 2 days.
  * Specimen Collections:
  * Collected at the same time as the NP specimen sent for COVID-19 testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: nasal pharyngeal (NP) swab samples — These donors will be from a population of patients who are already providing nasal pharyngeal (NP) swab samples in universal transport media (UTM) for COVID-19 testing at LabPMM LLC.
Diagnostic Test: peripheral blood draw — From patients suspected of SARS-CoV-2 viral infections.
  * At least 2mL to 5mL of peripheral blood.
  * Collected in EDTA tubes.
  * Shipped to ambient LabPMM, LLC within 2 days.
  * Specimen Collections:
  * Collected at the same time as the NP specimen sent for COVID-19 testing.
  * Collected two to three weeks post the original patient's COVID-19 testing.

SUMMARY:
Invivoscribe, Inc. and its wholly owned subsidiary LabPMM, LLC are collecting peripheral blood specimens from patients with suspected SARS-CoV-2 viral infections. These donors will be from a population of patients who are already providing nasal pharyngeal (NP) swab samples in universal transport media (UTM) for COVID-19 testing at LabPMM LLC. Specimens meeting this research protocol's inclusion criteria may be evaluated with various molecular techniques in order to identify nucleic acid sequences, antibodies, and/or antigens with the potential of being used to develop novel SARS-CoV-2 detection methods and COVID- 19 treatments and/or prevention methods (e.g. drug or vaccine development).

DETAILED DESCRIPTION:
This research protocol describes the collection and analysis of peripheral blood samples to:

* Identify nucleic acid sequences that may be used aide in the development of SARSCoV- 2 detection methods.
* Identify antibodies that may be used aide in the development of SARS-CoV-2 detection methods.
* Identify antigens that may be used aide in the development of SARS-CoV-2 detection methods. -Identify nucleic acid sequences that may be used aide in the development of COVID- 19 treatments and/or vaccines.
* Identify antibodies that may be used aide in the development of COVID-19 treatments and/or vaccines.
* Identify antigens that may be used aide in the development of COVID-19 treatments and/or vaccines.

ELIGIBILITY:
Inclusion Criteria:

* From patients suspected of SARS-CoV-2 viral infections.
* From patients who have had COVID-19 testing prescribed by their treating physicians.
* From patients whose COVID-19 test specimen was sent to LabPMM, LLC for testing

Exclusion Criteria:

* There are no exclusion criteria related to age, gender, race, ethnicity, geography, and/or other medical conditions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is an open study that will accept donations from any patients who both are being tested by LabPMM, LLC for COVID-19 and who sign the related ICF.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of nucleic acid sequencing, antibodies and antigens to be used in detection methods or treatments and/or vaccines | 2 years
  This research protocol describes the collection and analysis of peripheral blood samples to:
  * Identify nucleic acid sequences that may be used aide in the development of SARSCoV- 2 detection methods.
  * Identify antibodies that may be used aide in the development of SARS-CoV-2 detection methods.
  * Identify antigens that may be used aide in the development of SARS-CoV-2 detection methods.
  * Identify nucleic acid sequences that may be used aide in the development of COVID- 19 treatments and/or vaccines.
  * Identify antibodies that may be used aide in the development of COVID-19 treatments and/or vaccines.
  * Identify antigens that may be used aide in the development of COVID-19 treatments and/or vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: Jordon Thornes, Principal Investigator — Laboratory for Personalized Molecular Medicine,

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Company Website — http://invivoscribe.com